CLINICAL TRIAL: NCT01788605
Title: Prospective, Single-arm Phase 2 Trial to Evaluate Efficacy and Safety of Ramosetron in the Setting of Hematopoietic Stem Cell Transplantation for Hematologic Malignancies
Brief Title: Efficacy Study of Ramosetron in the Setting of Hematopoietic Stem Cell Transplantation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Ki-Seong Eom, MD, Associate Professor, The Catholic University of Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CBMTC-supp001
Record Dates: First submitted 2013-02-07; First posted 2013-02-11 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Hematologic Malignancies
Keywords: hematologic malignancies; hematopoietic stem cell transplantation; ramosetron; emesis
MeSH Terms: conditions — Hematologic Neoplasms; Vomiting | interventions — ramosetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ramosetron (Experimental)
  Interventions: Drug: ramosetron

INTERVENTIONS:
Drug: ramosetron

SUMMARY:
1. The purpose of this study is to determine the efficacy of ramosetron for the prevention of emesis and the control of nausea and vomiting despite of the prophylactic antiemetic treatment during hematopoietic stem cell transplantation
2. The study hypothesis is that ramosetron is effective for the prevention of emesis and control of emesis and/or vomiting that develop after the prophylactic antiemetic therapy in the setting of hematopoietic stem cell transplantation

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing hematopoietic stem cell transplantation conditioned with highly or moderately emetogenic drugs or total body irradiation (TBI) for hematologic malignancies
2. aged over 18 yrs
3. Eastern Cooperative Oncology Group (ECOG) performance status 0 - 2
4. patients who are able to take oral medications
5. patients who get well-informed and sign the consent

Exclusion Criteria:

1. Patients complicating

   * severe hypertension (systolic blood pressure > 210 mmHg or diastolic blood pressure > 120 mmHg)
   * significant heart disease such as congestive heart failure
   * renal insufficiency (serum Cr >= 3.0 mg/dL)
   * liver disease (Aspartate aminotransferase (AST), alanine aminotransferase (ALT) > 3 upper normal limit; alkaline phosphatase (ALP) > 2 upper normal limit)
2. Patients complicated by conditions such as gastrointestinal obstruction or active peptic ulcer causing emesis
3. Patients with brain tumor, brain metastasis and epilepsy
4. Patients with the history of extrapyramidal symptom
5. Patients with the history of allergy to serotonin antagonists
6. pregnant or lactating women
7. Patients with drug abuse or psychiatric illness, or patients who are not capable of the normal communications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2014-08; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
efficacy of ramosetron in terms of complete response (no emesis, no rescue therapy) during the conditioning regimen and within 3 or 6 days after the end of the conditioning regimen | within 1 week after the end of conditioning regimen

SECONDARY OUTCOMES:
the efficacy of second dose of ramosetron for the treatment of breakthrough emesis | within 1 week after the end of conditioning regimen

OTHER OUTCOMES:
the number of vomiting episodes | within 1 week after the end of conditioning regimen
grade of nausea and need for rescue therapy | within 1 week after the end of conditioning regimen

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic Blood & Marrow Transplantation Center, Seoul St Mary's Hospital, the Catholic University of Korea, Seoul, South Korea